CLINICAL TRIAL: NCT02875119
Title: A Phase 1 Trial to Evaluate the Safety, Pharmacokinetics (PK) and Pharmacodynamics (PD) of PC-6500 (Griffithsin [GRFT] in a Carrageenan Gel) in Healthy Women
Brief Title: Study to Evaluate the Safety of Griffithsin in a Carrageenan Gel in Healthy Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Population Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 728
Record Dates: First submitted 2016-08-15; First posted 2016-08-23 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Griffithsin Gel (Experimental): In the randomized period, duration of treatment will be 14 days; each of the 30 subjects will self-administer Griffithsin Gel once daily for 14 consecutive days, with 5 doses administered under clinical supervision and the remaining 9 doses administered at home.
  Interventions: Drug: Griffithsin Gel
- Placebo Gel (Placebo Comparator): In the randomized period, duration of treatment will be 14 days; each of the 30 subjects will self-administer placebo gel once daily for 14 consecutive days, with 5 doses administered under clinical supervision and the remaining 9 doses administered at home.
  Interventions: Drug: Placebo Gel

INTERVENTIONS:
Drug: Griffithsin Gel — Griffithsin Gel is a large biologic molecule that is intended for vaginal rather than systemic administration. In addition, Griffithsin Gel is being developed for the prevention of HIV infection and not as a therapeutic agent. The concentration of Griffithsin Gel associated with prevention of HIV in vitro and in vivo has been established in non-clinical studies (see Section 5). Studies have demonstrated that Griffithsin Gel is highly potent for HIV prevention and is effective at very low concentrations.
  One 4 mL dose of PC-6500, designed to provide an adequate vaginal concentration of GRFT for the prevention of HIV, based on preclinical data, will be evaluated. Rising dose tolerance is not the goal of this study because GRFT is likely to be minimally absorbed systemically, if at all.
  Arms: Griffithsin Gel
Drug: Placebo Gel — Placebo Gel
  Arms: Placebo Gel

SUMMARY:
This is a two-part study. The first part is a single-dose open label design. The second part employs a multiple dose, randomized, placebo controlled study design. Studies have demonstrated that GRFT is highly potent for HIV prevention and is effective at very low concentrations. One 4 mL dose of PC-6500, designed to provide an adequate vaginal concentration of GRFT for the prevention of HIV, based on preclinical data, will be evaluated. Rising dose tolerance is not the goal of this study because GRFT is likely to be minimally absorbed systemically, if at all.

ELIGIBILITY:
Inclusion Criteria:

* 1) Between 18 and 49 years of age (at screening), inclusive.
* 2) Willing and able to provide written informed consent.
* 3) Healthy, based on medical history, vital signs, physical examination, urinalysis, laboratory evaluations for genital infections and laboratory evaluations for hematology, liver and renal function.
* 4) HIV-negative as determined by HIV ELISA test at screening.
* 5) In the absence of the use of exogenous hormone(s), have a self-reported regular menstrual cycle, defined as having a minimum of 21 days and a maximum of 35 days between menses.
* 6) Normal Pap test at screening. (Documentation of normal Pap test results within 12 months prior to screening is also acceptable.)
* 7) Agrees to use effective contraception for the duration of the trial. If hormonal contraception or intrauterine device (IUD)/ Intrauterine system (IUS) is being used, it must be have been used for at least 30 days prior to screening, with no planned change in method during the study. The following forms of contraception (per self-report) are permitted: same-sex relationship, male or female sterilization, oral contraceptives, contraceptive implant, contraceptive patch, IUS, IUD depo-medroxyprogesterone acetate (DMPA; Depo-Provera®).
* 8) Willing to abstain from sexual intercourse/activity including receptive vaginal, oral, digital, and anal intercourse, and the use of any vaginal products including tampons, male and female condoms, contraceptive sponges, diaphragms, cervical caps, douches, lubricants, and vibrators/dildos; starting the Screening Visit (Visit 0) through the final safety visit (Visit 3/Day 8) in the OL period; and starting 48 hours before enrollment through the final safety visit (Visit 8/Day 21) in the randomized period
* 9) Agrees to not participate in any other clinical research for the duration of this trial.

Exclusion Criteria:

* 1) History of or known sensitivity/allergy to any component of either study product.
* 2) Currently pregnant or breast-feeding, or within 3 months of last pregnancy outcome.
* 3) Participation in any other clinical research trial involving investigational or marketed products currently or within two months of participation prior to screening, including any trial of a spermicide, microbicide and/or drug.
* 4) Known bleeding disorder that could lead to prolonged or continuous bleeding with biopsy.
* 5) Diagnosed with or treated for any STI or pelvic inflammatory disease in the last 3 months. Note: Women with a history of condylomata or genital herpes who have been asymptomatic for at least six months may be considered for eligibility.
* 6) Positive test for Neisseria gonorrhea (NG), Chlamydia trachomatis (CT), or Trichomonas vaginalis (TV) at screening.
* 7) Symptomatic vulvovaginal candidiasis, bacterial vaginosis (BV), or urinary tract infection (UTI) at screening. (Participants who test positive at initial screening may be treated and re-tested once, and reconsidered for screening).
* 8) Presence of any clinically significant genital epithelial findings (e.g. abrasions, ulcerations, or lacerations, or vesicles) suspicious for STIs at screening.
* 9) History of hysterectomy or menopause.
* 10) Use of excluded contraceptive methods including Nuvaring®, condoms (male or female), contraceptive sponge, diaphragm, or cervical cap.
* 11) History of gynecological surgery or procedure within past 2 months.
* 12) History of uterine prolapse, undiagnosed vaginal bleeding or urethral obstruction within the last 3 months, including unexplained break-through bleeding requiring sanitary protection.
* 13) Known current drug abuse, including illicit drugs, or alcohol abuse.
* 14) Abnormal finding on laboratory or physical examination or a social or medical condition which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of data.
* 15) Unable to comply with study requirements, including but not limited to, attending all study visits, using the gel as directed, observing abstinence throughout the study and use of allowable effective contraceptives.
* 16) History of latex allergy.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Number and percent of participants with TEAEs, SAEs and AEs leading to premature discontinuation. | 10 months
  To evaluate the safety of PC-6500 gel used vaginally for a single dose; and then for 14 consecutive days of dosing. AEs will be coded in accordance with the current version of the Medical Dictionary for Regulatory Activities (MedDRA).

SECONDARY OUTCOMES:
Evaluation of the area under the time-concentration curve of Griffithsin gel in blood during and after dosing as assessed by (AUC0-last; AUC0-∞) | 10 months
  To determine the PK of Griffithsin Gel in blood after a single dose, and then after 14 days of dosing.

CONTACTS AND LOCATIONS:
Overall Officials: George Creasy, MD, Study Chair — Population Council
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teleshova N, Keller MJ, Fernandez Romero JA, Friedland BA, Creasy GW, Plagianos MG, Ray L, Barnable P, Kizima L, Rodriguez A, Cornejal N, Melo C, Cruz Rodriguez G, Mukhopadhyay S, Calenda G, Sinkar SU, Bonnaire T, Wesenberg A, Zhang S, Kleinbeck K, Palmer K, Alami M, O'Keefe BR, Gillevet P, Hur H, Liang Y, Santone G, Fichorova RN, Kalir T, Zydowsky TM. Results of a phase 1, randomized, placebo-controlled first-in-human trial of griffithsin formulated in a carrageenan vaginal gel. PLoS One. 2022 Jan 20;17(1):e0261775. doi: 10.1371/journal.pone.0261775. eCollection 2022. PMID 35051209
- [Derived] Shrivastava-Ranjan P, Lo MK, Chatterjee P, Flint M, Nichol ST, Montgomery JM, O'Keefe BR, Spiropoulou CF. Hantavirus Infection Is Inhibited by Griffithsin in Cell Culture. Front Cell Infect Microbiol. 2020 Nov 4;10:561502. doi: 10.3389/fcimb.2020.561502. eCollection 2020. PMID 33251157